CLINICAL TRIAL: NCT05551949
Title: Mechanisms of Successful Vaginal Estrogen Prophylaxis for Postmenopausal Women With Recurrent Urinary Tract Infections: Urogenital Microbiota and Host Immune Responses
Brief Title: Preventing Recurrent UTI With Vaginal Estrogen
Acronym: PRUVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00314740; R01DK130856 (NIH)
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Urinary Tract Infection; Urinary Tract Infections; Cystitis Recurrent
Keywords: women
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Open label, single group clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaginal estrogen therapy (Other): Participants receive Vaginal estrogen therapy.
  Interventions: Drug: Vaginal estradiol tablets

INTERVENTIONS:
Drug: Vaginal estradiol tablets — Vaginal estradiol tablets (10mcg).

SUMMARY:
Among postmenopausal women who suffer from recurrent urinary tract infections (UTI), vaginal estrogen therapy prevents UTI recurrences for 50% of sufferers. This research will investigate why some women benefit but others do not, focusing on (a) the effects of vaginal estrogen therapy on the bacteria that inhabit the vagina and bladder, (b) its influence on immune responses in both compartments, and (c) the extent to which those changes are critical to successful UTI prevention. The findings will be a first step in the development of more effective strategies to prevent UTI, one of the most common and costly benign urologic conditions.

DETAILED DESCRIPTION:
Recurrent urinary tract infections (rUTI) are a significant problem among older women: 13% of female Medicare beneficiaries experience at least one UTI annually and >40% of these develop chronic recurrent UTI. Although UTIs are significantly reduced by vaginal estrogen therapy (VET), 50% of those using VET continue to experience UTI recurrences. It is unknown why some women benefit from VET while others do not. This application focuses on interrogating two mechanisms likely to be central to the effectiveness of VET. The first is the urogenital microbiota: an increase in vaginal lactobacilli is the purported mechanism by which VET reduces rUTI. Important and unanswered questions include how VET influences specific Lactobacillus spp., whether changes to specific Lactobacillus spp are the key to successful prophylaxis, and how VET affects the urinary microbiota. A second mechanism addressed by this application is the host vaginal and urinary immune response. Estrogen appears to influence localized urogenital immune responses, including Th17 and Th1 versus Th2 pathway signaling. Animal studies suggest that these compartmentalized immune responses play a critical role in UTI susceptibility, but human data are lacking. This application will address these unanswered questions. Postmenopausal women with rUTI will be treated with VET. Samples collected before and after VET will characterize vaginal and urinary microbiota, soluble mediators of inflammation in both compartments, and vaginal D-lactic acid. Aims 1 and 2 of this proposal will investigate the impact of VET on the urogenital microbiota and urogenital immune responses, respectively. Aim 3 will characterize the urogenital environments of participants who continue to experience rUTI during VET versus those who remain UTI-free. The accomplishment of these aims will provide pilot data for a larger and more definitive clinical trial. These proposed studies are a key step toward the investigators' goals of identifying biomarkers that reliably predict a successful response to rUTI prophylaxis and ascertaining the biological conditions required for successful UTI prevention. Ultimately, an understanding of the mechanisms of rUTI prevention will allow the development of novel and effective prevention strategies for postmenopausal women suffering from rUTI.

ELIGIBILITY:
Inclusion Criteria:

Participants in this study will be

* Postmenopausal women (menopausal for at least 1 year)
* Minimum age of 55 years
* Participants will have documentation of recurrent UTI, defined as follows:

  * History of treatment for at least 3 UTIs in the past year or 2 episodes within 6 months AND
  * At least one positive urine culture during an acute symptomatic episode.

Exclusion Criteria:

* Women receiving antibiotic prophylaxis to prevent UTI recurrence;
* Women with contraindications to vaginal estrogen (as indicated on the FDA-mandated package insert) and those who have used vaginal or systemic estrogen within the past 6 months;
* Women with an active UTI and those who have received antibiotics within the prior 2 weeks;
* Women with complicated rUTI, defined by immune compromise, anatomic or functional abnormalities of the urinary tract, indwelling catheterization, those performing self-catheterization, and those with neurological disease or illness relevant to the lower urinary tract;
* Women with only asymptomatic bacteriuria (rather than recurrent symptomatic UTI)

Ages: 55 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — identify as female
Enrollment: 27 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Vaginal microbiota | Baseline and 12 weeks
  Changes to relative vaginal abundance of key Lactobacillus spp. before and after treatment.
Change in Vaginal Interleukin-6 level | Baseline and 12 weeks
  Changes to vaginal Interleukin-6 before and after treatment.
Change in Urinary microbiota | Baseline and 12 weeks
  Changes to relative urinary abundance of key Lactobacillus spp. before and after treatment.
Change in Urinary Interleukin-6 level | Baseline and 12 weeks
  Changes to urinary Interleukin-6 before and after treatment.

SECONDARY OUTCOMES:
Urinary tract infection recurrence | Weeks 12 to 24
  Occurrence of symptomatic UTI after at least 12 weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Handa, MD MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after study completion
Supporting Information: Study Protocol, CSR
Time Frame: Data sharing will be provided within one year of study conclusion.
Access Criteria: To be determined